CLINICAL TRIAL: NCT03497078
Title: Comparison of Image Quality Between New Collimator LEHRS (General Electric - GE Healthcare) vs Siemens LEHR on Bone Scintigraphy
Brief Title: Comparison of Image Quality Between New Collimator LEHRS vs Siemens LEHR on Bone Scintigraphy
Acronym: LEHRS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHRO-2018-03
Record Dates: First submitted 2018-04-06; First posted 2018-04-13 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Comparison of Two Collimators During Bone Scintigraphy
Keywords: collimator; bone scintigraphy; image quality; scintigraphy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Refered patients for scintigraphy (Other)
  Interventions: Other: Bone scintigraphy

INTERVENTIONS:
Other: Bone scintigraphy — Comparison of image quality between new collimator LEHRS (General Electric - GE Healthcare) vs Siemens LEHR on bone scintigraphy.

SUMMARY:
Comparison of quality image with a new LEHRS GE collimator vs standard LEHR Siemens collimator on bone scintigraphy.

ELIGIBILITY:
Inclusion Criteria:

* Refered patients for scintigraphy

Exclusion Criteria:

* Under 18 y. old patients
* Pregnancy or supposed to be pregnant patients
* Kidney failure
* Painful patients
* Patients under guardianship
* Patients in whom a standard exam is not feasible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2018-04-03 (Actual); Primary Completion 2019-03-18 (Actual); Study Completion 2019-03-18 (Actual)

PRIMARY OUTCOMES:
visual quality of bone exams | Day 0

SECONDARY OUTCOMES:
Quantitative signal-noise-ratios | Day 0
quantitative datas on phantom | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Gilles METRARD, Dr, Principal Investigator — CHR d'Orléans
Locations (1):
- CHR d'Orléans, Orléans, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gilland DR, Welch BL, Lee S, Kross B, Weisenberger AG. Evaluation of a novel collimator for molecular breast tomosynthesis. Med Phys. 2017 Nov;44(11):5740-5748. doi: 10.1002/mp.12564. Epub 2017 Oct 13. PMID 28877351
- [Background] Songy B, Lussato D, Guernou M, Queneau M, Geronazzo R. Comparison of myocardial perfusion imaging using thallium-201 between a new cadmium-zinc-telluride cardiac camera and a conventional SPECT camera. Clin Nucl Med. 2011 Sep;36(9):776-80. doi: 10.1097/RLU.0b013e31821a294e. PMID 21825848